CLINICAL TRIAL: NCT02782663
Title: A Phase 2, Multicenter, Open-Label Extension (OLE) Study to Observe the Long-Term Efficacy, Safety, and Tolerability of Repeated Administration of Upadacitinib (ABT-494) in Subjects With Crohn's Disease
Brief Title: A Study to Evaluate the Long-Term Efficacy, Safety, and Tolerability of Repeated Administration of Upadacitinib (ABT-494) in Participants With Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-327; 2015-003759-23 (EudraCT Number)
Record Dates: First submitted 2016-05-23; First posted 2016-05-25 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Crohn's Disease (CD)
Keywords: Crohn's Disease; Efficacy; Safety; Tolerability; ABT-494
MeSH Terms: conditions — Crohn Disease | interventions — upadacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upadacitinib (ABT-494) Dose A (Experimental): Open label dose A once daily (QD)
  Interventions: Drug: ABT-494
- Upadacitinib (ABT-494) Dose B (Experimental): Open label dose B QD
  Interventions: Drug: ABT-494

INTERVENTIONS:
Drug: ABT-494 — Tablet: Oral
  Other Names: Upadacitinib; RINVOQ

SUMMARY:
This is a open-label extension (OLE) study designed to evaluate the long-term efficacy, safety, and tolerability of Upadacitinib (ABT-494).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have completed Study M13-740 through Week 52.
* If female, participant must be postmenopausal, surgically sterile or on using a birth control method.

Exclusion Criteria:

* For any reason participant is considered by the investigator to be an unsuitable candidate
* Female participant with a positive pregnancy test at Baseline or who is considering becoming pregnant during the study.
* Participant is not in compliance with prior and concomitant medication requirements and procedures throughout Study M13-740.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Remission | Up to Month 96
  It is defined as the percentage of participants achieving clinical remission and endoscopic remission.
Percentage of Participants in Remission at Week 0 Who Maintain Remission | Up to Month 96
  Remission is defined as participants achieving clinical remission and endoscopic remission.
Percentage of Participants Achieving Response | Up to Month 96
  It is defined as the percentage of participants achieving clinical response and endoscopic response.
Percentage of Participants Achieving Clinical Remission | Up to Month 96
  Clinical remission is defined based on the patient reported outcomes: average daily stool frequency and average daily abdominal pain.
Percentage of Participants Achieving Modified Clinical Remission | Up to Month 96
  Clinical remission is defined as change from baseline in the patient reported outcomes: average daily stool frequency and average daily abdominal pain.
Percentage of Participants Achieving Enhanced Clinical Response | Up to Month 96
  Enhanced clinical response is defined as change from baseline in the patient reported outcomes: average daily stool frequency and average daily abdominal pain.
Percentage of Participants Achieving Clinical Response | Up to Month 96
  Clinical response is defined as change from baseline in the patient reported outcomes: average daily stool frequency and average daily abdominal pain.
Percentage of Participants Achieving Endoscopic Remission | Up to Month 96
  Endoscopic remission is based on Simplified Endoscopic Score for Crohn's disease.
Percentage of Participants in Endoscopic Remission at Week 0 Who Maintain Endoscopic Remission | Up to Month 96
  Endoscopic remission is based on Simplified Endoscopic Score for Crohn's disease.
Percentage of Participants Achieving Endoscopic Improvement | Up to Month 96
  Endoscopic improvement is based on changes from baseline on the Simplified Endoscopic Score for Crohn's disease or endoscopic remission.
Percentage of Participants Achieving Endoscopic Response | Up to Month 96
  Endoscopic response is based on changes from baseline on the Simplified Endoscopic Score for Crohn's disease.
Percentage of Participants Achieving Crohn's Disease Activity Index (CDAI) Remission | Up to Month 96
  It is defined as CDAI less than 150.
Percentage of Participants Achieving Crohn's Disease Activity Index (CDAI) Response | Up to Month 96
  CDAI response is defined as a reduction in CDAI by >= 70 from baseline of Study M13-740.
Percentage of Participants Achieving Enhanced CDAI Response | Up to Month 96
  Enhanced CDAI response is defined as reduction in CDAI by >= 100 from baseline of Study M13-740.
Percentage of Participants Achieving Inflammatory Bowel Disease Questionnaire (IBDQ) Remission | Up to Month 96
  IBDQ remission is defined as IBDQ >= 170.
Percentage of Participants Achieving IBDQ Response | Up to Month 96
  IBDQ response is defined as an increase in IBDQ score >= 16 point from Baseline of Study M13-740.
Percentage of Participants Taking Steroids at Baseline (of Study M13-740) Who Are Steroid-Free | Up to Month 96
  Percentage of participants taking steroids at Baseline (of Study M13-740) who are steroid-free
Percentage of Participants Taking Steroids at Baseline (of Study M13-740) Who Are Steroid-Free for At Least 90 Days and Achieve Remission | Up to Month 96
  Percentage of participants taking steroids at Baseline (of Study M13-740) who are steroid-free for at least 90 days over time and achieve Remission
Percentage of Participants Achieving Remission and Normal C-Reactive Protein | Up to Month 96
  Percentage of participants achieving Remission and normal C-reactive protein. Remission is defined as Clinical Remission AND Endoscopic Remission.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (61):
- United States (27):
  - UC San Diego Health System /ID# 150041, La Jolla, California
  - Univ California, San Francisco /ID# 149987, San Francisco, California
  - Duplicate_University of Florida - Archer /ID# 150033, Gainesville, Florida
  - The Ctr for Gastro Disorders /ID# 150012, Hollywood, Florida
  - Nature Coast Clinical Research - Inverness /ID# 149975, Inverness, Florida
  - Gastroenterology Associates of Central Georgia, LLC /ID# 149870, Macon, Georgia
  - GI Specialists of GA, PC /ID# 150015, Marietta, Georgia
  - Cotton O'Neil Clinical Research Center, Digestive Health /ID# 149900, Topeka, Kansas
  - Duplicate_University of Louisville /ID# 149884, Louisville, Kentucky
  - Investigative Clinical Research /ID# 149886, Annapolis, Maryland
  - Charm City Research Group /ID# 150040, Towson, Maryland
  - Clin Res Inst of Michigan, LLC /ID# 150008, Chesterfield, Michigan
  - Mayo Clinic - Rochester /ID# 149894, Rochester, Minnesota
  - Kansas City Research Institute /ID# 149888, Kansas City, Missouri
  - Washington University-School of Medicine /ID# 149899, St Louis, Missouri
  - NYU Langone Long Island Clinical Research Associates /ID# 149976, Lake Success, New York
  - Weill Cornell Medicine/NYP /ID# 149895, New York, New York
  - Univ NC Chapel Hill /ID# 149982, Chapel Hill, North Carolina
  - University Of Cincinnati Medical Center /ID# 149977, Cincinnati, Ohio
  - Options Health Research, LLC /ID# 150010, Tulsa, Oklahoma
  - Texas Digestive Disease Consultants - Southlake /ID# 149869, Southlake, Texas
  - Texas Digestive Disease Consultants - Southlake /ID# 149989, Southlake, Texas
  - Aspen Clinical Research /ID# 150020, Orem, Utah
  - University of Virginia /ID# 149881, Charlottesville, Virginia
  - Virginia Mason Hospital & Medical Center /ID# 150042, Seattle, Washington
  - University of Washington /ID# 149988, Seattle, Washington
  - Wisconsin Center for Advanced Research /ID# 149863, Milwaukee, Wisconsin
- Duplicate_CHU de Liege /ID# 149912, Liège, Belgium
- Canada (5):
  - University of Alberta Hospital /ID# 149873, Edmonton, Alberta
  - University of British Columbia (UBC) - Gordon and Leslie Diamond Health Care Ce /ID# 149876, Vancouver, British Columbia
  - Duplicate_(G.I.R.I.) GI Research Institute Foundation /ID# 149878, Vancouver, British Columbia
  - Toronto Digestive Disease Associates /ID# 149877, Vaughan, Ontario
  - Disc_Royal Victoria Hospital / McGill University Health Centre /ID# 149871, Montreal, Quebec
- Hepato-Gastroenterologie HK, s.r.o. /ID# 149882, Hradec Králové, Czechia
- Denmark (2):
  - Kobenhavns Universitet - Hvidovre Hospital (HH) /ID# 149890, Hvidovre, Capital Region
  - Duplicate_Aarhus University Hospital /ID# 149919, Aarhus N, Central Jutland
- France (3):
  - CHRU Nancy - Hopitaux de Brabois /ID# 149896, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHRU Lille - Hopital Claude Huriez /ID# 149897, Lille, Nord
  - CHU Amiens-Picardie Site Sud /ID# 149921, Amiens, Somme
- Germany (3):
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 149936, Kiel, Schleswig-Holstein
  - DRK Kliniken Berlin Westend /ID# 149905, Berlin
  - Medizinisches Versorgungszentrum Portal 10 /ID# 149930, Münster
- Magyar Elhizastudomanyi Kozpont Kft. /ID# 149907, Budapest, Hungary
- Israel (3):
  - Yitzhak Shamir Medical Center /ID# 149943, Ẕerifin, Central District
  - The Chaim Sheba Medical Center /ID# 149945, Ramat Gan, Tel Aviv
  - Rabin Medical Center /ID# 149942, Petah Tikva
- Italy (2):
  - University of Catanzaro /ID# 149927, Catanzaro, Calabria
  - Duplicate_IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 149958, Bologna, Emilia-Romagna
- Netherlands (2):
  - Amsterdam UMC, locatie AMC /ID# 149932, Amsterdam, North Holland
  - Universitair Medisch Centrum Utrecht /ID# 149933, Utrecht
- Dunedin Hospital /ID# 149964, Otago, Otago, New Zealand
- Lovisenberg Diakonale Sykehus /ID# 149967, Oslo, Norway
- Poland (2):
  - Panstwowy Instytut Medyczny MSWiA w Warszawie /ID# 149978, Warsaw, Masovian Voivodeship
  - Santa Sp. z o.o. Santa Familia Centrum Badan, Profilaktyki i Leczenia /ID# 149979, Lodz, Łódź Voivodeship
- Cabinet Particular Policlinic Algomed /ID# 149993, Timișoara, Romania
- Slovakia (2):
  - Duplicate_KM Management, spol. s.r.o. /ID# 149949, Nitra, Nitra Region
  - Gastro I., s.r.o. /ID# 149948, Prešov, Presov
- Spain (2):
  - Hospital Arquitecto Marcide - Complejo Hospitalario Universitario de Ferrol /ID# 149996, Ferrol, A Coruna
  - Hospital Universitario La Paz /ID# 149997, Madrid
- United Kingdom (2):
  - Oxford University Hospitals NHS Foundation Trust /ID# 149963, Oxford, Oxfordshire
  - Duplicate_Manchester University NHS Foundation Trust /ID# 150006, Manchester

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] D'Haens G, Panes J, Louis E, Lacerda A, Zhou Q, Liu J, Loftus EV Jr. Upadacitinib Was Efficacious and Well-tolerated Over 30 Months in Patients With Crohn's Disease in the CELEST Extension Study. Clin Gastroenterol Hepatol. 2022 Oct;20(10):2337-2346.e3. doi: 10.1016/j.cgh.2021.12.030. Epub 2021 Dec 27. PMID 34968730
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/